CLINICAL TRIAL: NCT01061918
Title: Evaluation Of Bilateral Tecnis Multifocal Versus ReSTOR 3D Intraocular Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: William Lahners, Center For Sight
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: Tecnis MF/Restor
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Cataract
Keywords: Compare the visual outcomes with bilateral implantation of Tecnis MF and ReSTOR IOLs 6 months post cataract surgery.
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tecnis MF (Active Comparator)
  Interventions: Device: Tecnis MF
- ReSTOR (Active Comparator)
  Interventions: Device: ReSTOR

INTERVENTIONS:
Device: Tecnis MF — 20 patients in the Tecnis MF group.
  Arms: Tecnis MF
Device: ReSTOR — 20 patients in the ReSTOR group.
  Arms: ReSTOR

SUMMARY:
The purpose of this study is to compare the visual outcomes with bilateral implantation of Tecnis MF and ReSTOR intraocular lenses (IOLs) 6 months post cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation has been planned for both eyes
* Visual potential of 20/30 or better in each eye after cataract removal and IOL implantation
* Preoperative best-corrected distance visual acuity (BSDVA) worse than 20/40 Snellen. If there is a glare component, glare testing which reduces the visual acuity to less than 20/40
* Naturally dilated pupil size (in dim light) > 3.5 mm (with no dilation medications) for both eyes
* Preoperative corneal astigmatism of 1.0 D or less
* Clear intraocular media other than cataract
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Use of systemic or ocular medications that may affect vision
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus, immunocompromised, etc.)
* Subjects with diabetes mellitus
* Uncontrolled systemic or ocular disease
* History of ocular trauma or prior ocular surgery
* Amblyopia or strabismus
* Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 4.0 mm under mesopic/scotopic conditions)
* Contact lens usage within 6 months for polymethyl methacrylate (PMMA) contacts lenses, 1 month for gas permeable lenses or 1 week for extended-wear and daily-wear soft contact lenses
* Requiring an intraocular lens <15.0 or >26.0 diopters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Refraction | 1 year
Distance Visual Acuities | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - William Trattler, Miami, Florida
  - William Lahners, Sarasota, Florida